CLINICAL TRIAL: NCT03511833
Title: Comparison of Treatment by IN Ketamine to IV Morphine in Acute Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, michal roll, Director, R&D Department, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TASMC-18-PH-0459-17-CTIL
Record Dates: First submitted 2018-03-05; First posted 2018-04-30 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Acute Traumatic Pain
Keywords: Intra nasal ketamine; IV morphine; acute traumatic pain
MeSH Terms: interventions — Morphine; Ketamine

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized according to a blocked randomization scheme using www.sealedenvelope.com (site accessed Sep 10, 2017), which permits assignment of the participant to either group "A" or "group B" (the IN ketamine or IV morphine group). Only the pharmacy will have knowledge of which group is Ketamine and which group is Morphine. Eligible patients will be divided in equal proportions (58 in group A and 58 in group B). Both medications will be prepared by the pharmacy as coded kits, and will be stored in the ER safe with clear signage: "For ketamine/morphine clinical trial only". Shelf life of the kits is 6 months. Each vial in a kit will be marked by the group name either "A" or "B" and by either "IN" or "IV". The "IV" vials will either contain: morphine (10 mg of morphine in 10 ml saline) or 10 ml saline for IV administration, and the "IN" vials will either contain ketamine (100 mg in 2ml saline) or 2 ml saline for nasal administration.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morphine group (Active Comparator): Morphine group will receive IV medication and IN saline.
  Interventions: Drug: Morphine
- Ketamine group (Experimental): Ketamine group will receive IV saline and IN medication.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Morphine — IV morphine -0.1 mg/kg: Morphine vial contains 10 mg/10 ml = 1mg/ml ----> 0.1 ml/kg
  Other Names: no other Intervention name
  Arms: Morphine group
Drug: Ketamine — IN ketamine: 1 mg/kg: Ketamine vial contains 100 mg/2 ml = 50mg/ml ---> 0.02ml/kg
  Other Names: no other Intervention name
  Arms: Ketamine group

SUMMARY:
Patients who present with acute traumatic injuries in the pre-hospital setting or to the emergency department (ED) are treated with opioids, the current gold standard for severe acute pain therapy. Treatment with opioids has many disadvantages: the need of skilled manpower to administer the medication IV, numerous side effects- mainly cardiorespiratory depression- which necessitates post medication administration continuous monitoring of patients. IV administration may be difficult or impossible to provide in a number of extreme circumstances. For these reasons, there is a constant search for alternate treatment options for pain in acute traumatic injuries. IN ketamine has only recently been studied favorably in our department in adults, in an open, prospective study (Shimonovich at al 2016), and warrants further investigation in the setting of acute traumatic pain. Ketamine is a safe and efficacious analgesic and is overall well received both by patients and physicians. Side effects include: hallucinations and dissociation. As opposed to opioids, ketamine does not alter patients' respiratory and hemodynamic stability giving ketamine great therapeutic potential for pain reduction in trauma patients, pre-hospital patients, and battlefield injuries. The study we are conducting is designed to test and analyze the safety and efficacy of IN Ketamine compared to IV morphine in a setting of acute traumatic pain in the ED, when both medications are administered by the protocol as is customary for treatment of pain in the Emergency Medicine department, and will be a prospective, randomized, double blind, controlled study.

DETAILED DESCRIPTION:
The procedure:

1. Eligible patients will be identified by the ED personnel. They will make sure to inquire about and also visually inspect the patient's nares regarding nasal congestion, deviated septum, obstruction or injury.
2. Research physician will address the patient, explain about the trial and ask the patient to sign a consent form.
3. The patient will be randomized and assigned to a trial group: "A" or "B" and it will be noted in the Data sheet.
4. According to physician order (IV amount and IN amount) and patient group assignment, the nurse will prepare two blinded syringes that will be marked "A" or "B" (the assigned group) and "IN" or "IV" and note in the data sheet the time of syringe preparation.
5. The IV syringe will contain either Morphine or Normal Saline (up to 10 ml), and the IN syringe will contain either Ketamine or Normal saline (up to 2 ml).
6. The amount in the syringes will be calculated based on the patients' weight:

   IV-0.1 mg/kg: Morphine vial contains 10 mg/10 ml = 1mg/ml ----> 0.1 ml/kg IN-1 mg/kg: Ketamine vial contains 100 mg/2 ml = 50mg/ml ---> 0.02ml/kg
7. Administration of the medication is limited to one hour from preparation in the syringe.
8. The nurse will hand the syringes to the researcher (blinded and coded) and note in the data sheet the time of administration and the amount to administer IN and IV.
9. Prior to administering medication to the patient the researcher will measure vital signs (blood pressure, heart rate, respiratory rate, and O2 saturation) as well as pain level on a 100 mm VAS (visual analogue scale) questionnaire.
10. After administration of medications the researcher will measure vital signs (blood pressure, heart rate, respiratory rate, and O2 saturation) as well as pain level on a 100 mm VAS questionnaire every 5 minutes for the first 30 minutes and then every 15 minutes after that at 30, 45, 60, and 90 minutes.

    Saturation >95% on room air; if lower than 90%, the patient will be placed on 40% oxygen mask.
11. Measurement of vital signs will not interfere with any other treatment that the patients receives for their injury in the ED.
12. If the patient will be moved to another department from the ED, they will be withdrawn from the study.
13. Cardiorespiratory follow-up (as per bullet point number 8 above), will be concluded at 1.5 hours post-intervention, and clinical follow-up will continue as long as the patient remains in the ED.
14. 90 minutes after drug administration, if pain had not subsided sufficiently according to treating physician's clinical assessment, patient will receive further analgesic medications by physician order, as per ED protocol. The protocol takes into account concurrent medications (in this case either morphine or ketamine. Neither morphine nor ketamine will be used in these patients after test drug administration.

ELIGIBILITY:
Inclusion Criteria:

* be 18-70 years old
* self-report pain greater than or equal to 7/10 on a numerical-verbal scale
* weigh 50-100 kg
* have an ASA (American Society of Anaesthesiologists' classification) score of 1-2
* have systolic blood pressure of 90-160 mmHg

Exclusion Criteria:

* have had opioid analgesia administered within 2 hours of the study
* are chronic analgesia users (of opioid or others)
* have known allergies to morphine or ketamine
* have had a large meal within an hour prior to trauma
* are pregnant
* have a psychiatric history
* have nasal congestion, nasal trauma, epistaxis, or a deviated nasal septum
* have suffered any head or face trauma: any trauma that is manifested by an external mark in the face or skull.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of intranasal ketamine in decreasing pain intensity [patient assessed - VAS pain score] [ Time Frame: 2 hour post administration | 2 hours
  Time to achieve a clinically meaningful pain reduction was defined as the first time-point at which the patient reported 15mm of pain reduction or more. Maximal pain reduction was defined as the lowest VAS score reported by the patient over the course of follow-up. Time to maximal pain reduction was defined as the time at which the patient has the lowest VAS score over the course of the 2 hours follow-up.

SECONDARY OUTCOMES:
• adverse effects [Opiate Related Symptom Distress Scale] [ Time Frame: 2 hour post administration ] | 2 hours
  Adverse effects were recorded at the end of two hours using the 'Opiate Related Symptom Distress Scale' and included measurements of the presence, frequency, intensity and disruptiveness of 12 common opiate side-effects. Among these were nausea, vomiting, urinary retention, constipation, difficulty concentrating, dizziness, confusion, and others.
• patient satisfaction [Interview] [ Time Frame: 2 hours post administration ] | 2 hours post administration
  patients were asked to provide subjective comments

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, department of Emergency Medicine, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
a table summering pain assessing questioners will be available from corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP